CLINICAL TRIAL: NCT04368104
Title: Endometrial Changes and Fallopian Tubal Darwishscope Test (Office Hysteroscopic Bubble Suction and Tubal Peristalsis) in Women Using Progesterone-only Contraception (POC) as Noticed by Office Hysteroscopy.
Brief Title: Office Hysteroscopy in Women Using Progesterone-only Contraception (POC)
Status: Completed | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: Darwish test and POC
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fallopian Tube Peristalsis and Patency; Endometrial Pattern
Keywords: hysteroscopy; tubal patency; bubble suction test; tubal peristalsis; minipills; endometrium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: women using any form of minipills
  Interventions: Diagnostic Test: Darwish test (office hysteroscopic bubble suction and tubal peristalsis)
- Group B: women subjected to office hysteroscopy for different indications but not using any form of hormones or systemic or local hormonal contraception.
  Interventions: Diagnostic Test: Darwish test (office hysteroscopic bubble suction and tubal peristalsis)

INTERVENTIONS:
Diagnostic Test: Darwish test (office hysteroscopic bubble suction and tubal peristalsis) — Testing Darwish test (office hysteroscopic bubble suction test and proximal tubal peristalsis) in women using minipills versus other cases not using hormones..

SUMMARY:
Mechanisms of action of progesterone-only contraception (POC) include endometrial and Fallopian tubal changes without any scientific documentation. We succeeded to document proper assessment of the proximal part of the Fallopian tubes and test anatomic tubal patency as well (Darwishscope test) via hysteroscopy. This study will test endometrial pattern and Fallopian tubal status in women using progesterone-only contraception (POC) utilizing office hysteroscopy.

DETAILED DESCRIPTION:
progesterone-only contraception (POC) prevent pregnancy by thickening the mucus in the cervix to stop sperm reaching an egg and assumed to increase Fallopian tubal motility so the fertilized oocyte reaches the endometrial cavity too early for implantation. However, this assumption has no scientific documentation so far. We succeeded to document visualization of peristalsis of the proximal part of the Fallopian tubes and anatomic tubal patency as well (Darwish test) via hysteroscopy.

Aim of study: to evaluate endometrial pattern and Darwishoscope test (office hysteroscopic bubble suction test and proximal tubal peristalsis) in women using progesterone-only contraception (POC).

Intervention:

It will include women using any form of minipills (Desogestrel 75 µg, or Norethisterone 350 µg), medroxy-progesterone acetate, Merina or implanon complaining from abnormal uterine bleeding in the form of menorrhagia, metorrhagia, intermenstrual spotting or or postcoital bleeding. Cases with suspected endometrial lesion by routine transvaginal follow-up of those cases were also included. They will be assigned as group A. Group B will include women subjected to office hysteroscopy for different indications but not using any form of hormones or systemic or local hormonal contraception. Preoperative counseling of all patients followed by an informed written consent taken from those who will agree. The included patients subjected to complete history taking and meticulous physical examination. A suspected pregnancy, heavy vaginal bleeding, active pelvic inflammatory disease (PID), severe co-morbidity, e.g., severe cardiac, neurologic, or chest disease, and other medical contraindications to pregnancy will be exclusion criteria of this study. Selected cases will be subjected to office hysteroscopy.

Sample size calculation is based on our previous study on the prevalence of tubal peristalsis seen via hysteroscopy. If it is supposed that tubal peristalsis would be positive in about 40% of apparently normal FT and it would be positive in about 80% of cases taking progesterone-only contraception (POC), sample size in each group would be 73 cases in each group. This means 73 or more measurements/surveys are needed to have a confidence level of 90% that the real value is within ±5% of the measured/surveyed value ( α error of 0.05 (the real value is within ±5% of the measured/surveyed value). The vulva, vagina and the thighs will be disinfected with a 10% povidone-iodine solution. Sterile draping will be applied.

Office diagnostic hysteroscopy will be performed using a 2.6 mm 30° rigid scope with a 3.2mm outer sheath (Karl Storz, Tutlingen, Germany). At the beginning in all cases vaginoscopic approach is tried but if any difficulty will be encountered, grasping of the anterior lip of cervix with a volsellum will be done. Thereafter, the uterus will be distended with normal saline at 100-150 mmHg generated from a pneumatic cuff of sphygmomanometer wrapped around the 500-cm3 infusion bottle. As attached to a 250-W Xenon light source, the scope will be introduced gently through the cervical canal and internal os. To perfectly perform hysteroscopic Darwish test the following tricks should be followed. Clear view of the endometrial cavity should be achieved on panoramic view by placing the hysteroscope at internal os waiting for a while to achieve homogenous distension. The uterine cavity should be systematically examined starting by its anterior and posterior walls, the fundus, and the borders. Examination will be considered complete if the both tubal ostia will be reached describing any gross pathology, e.g., septum, adhesions, polyp(s), myoma, and any growth.

Prerequisites for a successful access to evaluate fallopian tubes via hysteroscopy include utilization of a 300 telescope with gaining skill of its rotation to reach both cornea and most importantly orientation with a fundamental anatomic triad (Darwish triad) (DT). The most proximal corneal fine wide circle is the ostium (the end of the endometrial cavity) representing a base of a cone which is followed by a shallow conical groove (the first millimeters of the intramural part of FT). Finally, a distal pinhole dark spot (the narrowest part of the FT) representing the tip of the cone. Putting DT (ostium, intramural part and dark spot) in mind is the key step to evaluate tubal patency and physiology via hysteroscopy. If DT is clearly accessible, the hysteroscopist should comment on this. If there are some osteal lesions like tiny polyp(s) or fine adhesions that may hinder proper evaluation of the tubal anatomy and physiology, the hysteroscopist should notice and document. Passage of any air bubbles in the irrigating fluid towards DT is reported. If no observed air bubbles, the hysteroscopist should inject just 2 ml of air into the rubber end of the sterile infusion set. Hysteroscopic bubble suction test is considered positive if air bubbles are sucked by DT within 1 min. During this period, neither injection of air nor increased pressure will be done. If no suction of gas bubbles occurred, the examiner should wait for 1 min more to exclude tubal spasm. Again, if no suction of the bubbles by DT and their accumulation at the corneal end, the test will be considered negative. Simultaneously, careful visualization of any change in the shape of the ostium and intramural part of FT particularly during suction of the air bubbles will be recorded in all cases. Tubal peristalsis is defined as observed osteal and intramural tubal rhythmic opening and closing on maintained intrauterine pressure, i.e., periodic changes of DT in the form of widening followed by collapse on meticulous observation. If the ostium and intramural part of the tube is obviously opened followed by collapse and non-visualization of the pinhole dark spot of DT for a while, positive peristalsis will be reported. The same steps will be repeated on the contralateral side and reported.

ELIGIBILITY:
Inclusion Criteria:

* women using progesterone-only contraception (POC)
* women planned for office hysteroscopy for other indication.

Exclusion Criteria:

* A suspected pregnancy.
* heavy vaginal bleeding.
* active pelvic inflammatory disease (PID).
* severe co-morbidity, e.g., severe cardiac, neurologic, or chest disease
* Other medical contraindications to pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women using any form of progesterone-only contraception (POC) including minipills (Desogestrel 75 µg, or Norethisterone 350 µg), MPA, Merina or Implanon asigned as group A and women subjected to office hysteroscopy for other indications (group B).
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
office hysteroscopic endometrial and Fallopian tubal Darwishscope test in women using progesterone-only contraception (POC) versus non users of any hormones.. | 1 month
  case control

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No